CLINICAL TRIAL: NCT05295368
Title: Strategies for Kidney Outcomes Prevention and Evaluation - The SKOPE Study
Acronym: SKOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Professor Tazeen Jafar, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CSASI20nov-0001
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; clinical trial; primary care; kidney function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multicomponent intervention (Experimental): 1) 1. Training Nurses/service coordinators as Health Coaches and Hybrid Follow-up Approach of in-person, Telephone and Secure Video Sessions; 2)Training physicians in algorithm-based standardized management of CKD and hybrid care delivery;3) subsidy on sodium-glucose transport protein-2 inhibitors (SGLT-2i) for CKD; and 4) regular CKD case review meetings.
  Interventions: Other: Multicomponent intervention
- Usual care (No Intervention): treated by physicians and nurses who are not trained in SKOPE treatment algorithms.

INTERVENTIONS:
Other: Multicomponent intervention — Intervention includes four components 1) training nurses as health coaches for motivational conversation and CKD specific lifestyle counseling on diet and exercise, using hybrid follow-up approach of in-person, telephone, and secure video sessions; 2)Training physicians in algorithm-based standardized management of CKD and hybrid care delivery;3) subsidy on sodium-glucose transport protein-2 inhibitors (SGLT-2i) for CKD; and 4) regular CKD case review meetings.
  Arms: multicomponent intervention

SUMMARY:
Background: Chronic kidney disease (CKD) is a major public health threat associated with significant morbidity, high mortality, and reduced quality of life. However, empirical evidence is limited on strategies to enhance the effectiveness of care for CKD. The objective of the trial is to evaluate the effectiveness and cost-effectiveness of multicomponent primary care strategies in preserving kidney function among patients with CKD at primary care clinics in Singapore.

Methods: A pragmatic, randomized controlled trial, in 4 socioeconomically diverse primary care clinics (polyclinics) in Singapore over 3 years. A total of 896 participants with CKD Stage 3 or worse aged ≥40 and <80 years will be enrolled, with 224 from each polyclinic. Participants enrolled in each polyclinic will be randomly allocated to the intervention or usual care group in a 1:1 ratio.

Intervention includes four components 1) training nurses as health coaches for motivational conversation and CKD specific lifestyle counseling on diet and exercise, using hybrid follow-up approach of in-person, telephone, and secure WhatsApp video meetings; 2)Training physicians in algorithm-based standardized management of CKD and hybrid care delivery;3) subsidy on sodium-glucose transport protein-2 inhibitors (SGLT-2i) for CKD; and 4) regular CKD case review meetings.

Patients in the usual care arm will be treated by physicians and nurses who and are not trained in SKOPE treatment algorithms.

Study outcomes:

The primary outcome will be the eGFR total slope from randomization to final follow-up at 36 months. secondary effectiveness outcomes will be 1) Change in CVD risk score as measured by The Million Hearts Longitudinal ASCVD Risk Assessment score 2) Change in CKD quality of life measured by KDQOL-36TM

ELIGIBILITY:
4.3 Inclusion Criteria

* Patients with CKD Stage 3 or Stage 4 defined as persistent reduction in Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula eGFR ≥15 and < 60 ml/min/1.73m2 for at least 3 months based on two eGFR readings at least 3 months apart and the last eGFR should be measured at least 3 months ago.
* Receiving care at the polyclinics in Singapore for at least one year at the time of recruitment
* Age >=40 and <80 years
* Singaporean or permanent resident

4.4 Exclusion Criteria

* On kidney replacement therapy
* Pregnancy or breastfeeding
* Known terminal illness
* Recent hospitalization during last 3 months
* History of leg or foot ulcers, severe mental illness, prior kidney transplant
* Inability to provide informed consent

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
the eGFR | from randomization to final follow-up at 36 months

SECONDARY OUTCOMES:
Mean change in CVD risk score | at 12, 24, and 36 months from the baseline
  measured by The Million Hearts Longitudinal atherosclerotic cardiovascular disease(ASCVD) Risk Assessment score:not assessed via a scale. Results are given as a percent (%) on a scale of less than 1% to 99.99%. A higher score indicates a higher risk
Mean change in CKD quality of life | at 12, 24, and 36 months from the baseline
  Assessed by Kidney Disease Quality of Life 36-item short form survey(KDQOL-36TM), score ranges from 0 to 100, higher scores dente better quality of life
Mean change in CKD quality of life | at 12, 24, and 36 months from the baseline
  Assessed by The 5-level EuroQol-5D version (EQ-5D-5L):Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).

OTHER OUTCOMES:
Incident eGFR <30 ml/min/1.73m2 | from randomization to final follow-up at 36 months
Incident eGFR <45 ml/min/1.73m2; | from randomization to final follow-up at 36 months
Incident eGFR <15 ml/min/1.73m2; | from randomization to final follow-up at 36 months
Incident ACR >300 mg/g; | from randomization to final follow-up at 36 months
Incident dialysis | from randomization to final follow-up at 36 months
Rate of MACE (composite of total death, myocardial infarction, coronary revascularization, stroke, and hospitalization because of heart failure | from randomization to final follow-up at 36 months
Mean change in kidney failure risk equation ( KFRE) score | from randomization to final follow-up at 36 months
  The score is based on an equation not on a scale,Results are given as a percent (%) on a scale of less than 1% to 99.99%. A higher score indicates a higher risk
Proportion of subjects who experienced albuminuria defined as ACR >30 mg/g | from randomization to final follow-up at 36 months
  defined as ACR >30 mg/g
Rate of All-cause mortality | from randomization to final follow-up at 36 months
Rate of CVD deaths | from randomization to final follow-up at 36 months
Rate of hospital admission due to CHD, heart failure, or stroke | from randomization to final follow-up at 36 months
Mean change in Dietary score | from randomization to final follow-up at 36 months
  Not based on a scale, higher score indicates better outcome
Mean change in level of physical activity | from randomization to final follow-up at 36 months
  International Physical Activity Questionnaire (PHAQ): there is no range, higher scores denote higher levels of physical activities
Mean change in BMI | from randomization to final follow-up at 36 months
Mean change in adherence to antihypertensive | from randomization to final follow-up at 36 months
Mean change in adherence to glucose-lowering medication | from randomization to final follow-up at 36 months
Mean change from baseline in therapeutic intensity score of antihypertensive medication (all and class specific) therapeutic intensity score (summary measure that accounts for the number of medications and the relative doses a patient received) | from randomization to final follow-up at 36 months
  summary measure that accounts for the number of medications and the relative doses a patient received. Higher scores indicate higher dose.
Mean change in Framingham risk score | from randomization to final follow-up at 36 months
  based on an equation, Results are given as a percent (%) on a scale of less than 1% to 99.99%. A higher score indicates a higher risk
Proportion of subjects with at least 40% decline in baseline eGFR or kidney replacement therapy ( KRT) with mortality | from randomization to final follow-up at 36 months
b) Proportion of subjects with at least 40% decline in baseline eGFR or KRT without mortality | from randomization to final follow-up at 36 months
c) Proportion of subjects with at least 50% decline in baseline eGFR or KRT with mortality | from randomization to final follow-up at 36 months
d) Proportion of subjects with at least 50% decline in baseline eGFR or KRT without mortality | from randomization to final follow-up at 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jafar TH, Tan NC, Gandhi M, Yoon S, Finkelstein E, Seng PMK, Ong R, Thiagarajah AG, Lee BL, To KC, Moosa AS. Evaluating a multicomponent intervention for managing kidney outcomes among patients with moderate or advanced chronic kidney disease (CKD): protocol for the Strategies for Kidney Outcomes Prevention and Evaluation (SKOPE) randomized controlled trial. Trials. 2024 Oct 30;25(1):730. doi: 10.1186/s13063-024-08564-1. PMID 39472975